CLINICAL TRIAL: NCT05713838
Title: Organ Preservation With Durvalumab-based Immunotherapy in Combination With Chemoradiation as Definitive Therapy for Early Stage, cT1 and cT2N0, Esophageal Adenocarcinoma With Indication for Radical Surgery: A Prospective, Multicenter Study of the FLOT-AIO Gastric Cancer Group
Brief Title: Organ Preservation With Durvalumab-based Immunotherapy in Combination With Chemoradiation as Definitive Therapy for Early Stage Esophageal Adenocarcinoma With Indication for Radical Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRESTO
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Esophagus Adenocarcinoma
Keywords: esophageal adenocarcinoma; GEJ adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Patients eligible for this trial will be enrolled into one of two cohorts:
  Cohort 1 will consist of participants with PD-L1 combined positive score (CPS) < 10.
  Cohort 2 will consist of participants with PD-L1 CPS ≥ 10.
  Patients in both cohorts will receive immunotherapy with durvalumab in parallel to 2 cycles FLOT chemotherapy induction followed by immunotherapy with durvalumab in parallel with 3 cycles of modified FOLFOX chemotherapy plus concomitant radiation (50 Gy).
  After initial core treatment and endoscopic re-evaluation patients with complete remission will receive durvalumab monotherapy (1500 mg, IV, Q4W) for a maximum of 12 cycles.
  Patients in whom a locoregional persistence is confirmed will be offered surgical resection instead of entering the the maintenance period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Chemoradiotherapy (Experimental): Core Treatment:
  * D1: Durvalumab (1500 mg, IV) PLUS FLOT (50 mg/m² docetaxel, 85 mg/m² oxaliplatin, 200 mg/m² calcium folinate and 2600 mg/m² 5-FU 24h)
  * D15: FLOT (50 mg/m² docetaxel, 85 mg/m² oxaliplatin, 200 mg/m² calcium folinate and 2600 mg/m² 5-FU 24h),
  * D29: Durvalumab (1500 mg, IV) PLUS mFOLFOX (85 mg/m² oxaliplatin, 200 mg/m² calcium folinate, 400 mg/m² 5-FU bolus and 1600 mg/m² 5-FU 48h) PLUS 50 Gy radiotherapy
    * 5 weeks with 5 days a week radiotherapy (25 daily fractions, 2.0 Gy = ∑50Gy)
  * D43: mFOLFOX (85 mg/m² oxaliplatin, 200 mg/m² calcium folinate, 400 mg/m² 5-FU bolus, 1600 mg/m² 5-FU 48h) (radiation cont.)
  * D57: Durvalumab (1500 mg, IV) PLUS mFOLFOX (85 mg/m² oxaliplatin, 200 mg/m² calcium folinate, 400 mg/m² 5-FU bolus and 1600 mg/m² 5-FU 48h) (radiation cont.)
  Maintenance Phase Durvalumab monotherapy max. 12 cycles à 4 weeks:
  Durvalumab (1500 mg, IV, Q4W) D1
  Interventions: Drug: Durvalumab; Drug: FLOT; Drug: mFOLFOX-6; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Durvalumab — 1500 mg Durvalumab, IV, day 1 Q4W (max. 15 cycles)
  Other Names: IMFINZI
Drug: FLOT — 50 mg/m² docetaxel, 85 mg/m² oxaliplatin, 200 mg/m² calcium folinate and 2600 mg/m² fluorouracil as 24 h-infusion, 2 cycles
Drug: mFOLFOX-6 — 85 mg/m² oxaliplatin, 200 mg/m² calcium folinate, 400 mg/m² fluorouracil as bolus dose and 1600 mg/m² fluorouracil as 48 h-infusion, ² cycles
Radiation: Radiotherapy — 5 weeks with 5 days a week radiotherapy (25 daily fractions with 2.0 Gy = ∑50Gy)

SUMMARY:
The present clinical trial is a prospective, investigator-initiated, single-arm, open-label, multicenter phase II trial investigating whether a definite organ preservation therapy consisting of the combination of durvalumab with chemoradiation is an efficient and safe treatment option for early stage, cT1 and cT2N0, esophageal adenocarcinoma with indication for radical surgery.

DETAILED DESCRIPTION:
Patients with early stage, cT1 and cT2N0 esophageal adenocarcinoma with indication for radical surgery (esophagectomy or transhiatal extended gastrectomy) will be enrolled in two cohorts according to their PD-L1 CPS (cohort 1 CPS < 10, cohort 2 CPS ≥ 10). All patients will receive core treatment consisting of immunotherapy with durvalumab in parallel to 2 cycles FLOT chemotherapy, followed by immunotherapy with durvalumab in parallel to 3 cycles of modified FOLFOX plus concomitant radiation (50 Gy). Eight weeks after this, patients will undergo tumor assessment consisting of esophagogastroduodenoscopy with extensive biopsies (bite-on-bite biopsies and fine-needle aspiration), endoscopic ultrasonography with measurement of maximum tumor thickness, and CT- or MRI-scans for tumor re-evaluation. Surgical resection would be offered only to those patients in whom a locoregional persistence is confirmed on tumor assessment, in the absence of any signs of distant dissemination. Patients with complete remission will enter the maintenance phase receiving durvalumab monotherapy for up to 12 cycles.

The primary objective of this trial is to investigate the treatment efficacy of the combination of durvalumab and chemoradiation as organ preservative treatment option avoiding mortality and surgical complications with rate of clinical and pathological complete response (cCR/pCR) at time of endoscopic re-evaluation defined as primary efficacy endpoint.

The secondary objectives are the further assessment of the efficacy of the combination of durvalumab and chemoradiation as organ preservative treatment option 1-/2- and 3-year cCR/pCR rate, rate of salvage surgery, 90-day and 1-year mortality as secondary endpoints and to assess the quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given written informed consent.
2. Patient is, in the investigator's judgement, willing and able to comply with the study protocol including the planned surgical treatment.
3. Patient is ≥ 18 years of age at time of signing the written informed consent.
4. Patient has been diagnosed with histologically confirmed esophageal adenocarcinoma (including gastroesophageal junction (GEJ) (Siewert I-III)) with:

   1. cT2 N0 M0 stage or T1 N0 M0 stage and a given indication for radical surgical resection to current S3-guidelines (this includes patients with a given indication for radical surgery after endoscopic-resection of a cT1-2 N0 M0 tumor [poor grading or L1/V1 invasion or basal R1 resection or deep submucosal infiltration]) (see section 4.2.3 for detailed information).
   2. tumor is considered medically and technically resectable.
5. Tumor is tested (local testing with validated assays is sufficient, e.g., Dako PD-L1 IHC 22C3 or 28-8) for PD-L1 according to combined positive score (CPS) and results must be available prior study enrollment. In addition, tumor should be tested locally for MSI status and PD-L1 according to tumor proportion score (TPS) OR a representative tumor specimen that is suitable for central determination of PD-L1 TPS and MSI status is available. The analysis requires paraffin embedded biopsy samples of the tumor to be provided to the Sponsor.

   NOTE: It is encouraged that CPS, TPS and MSI testing is performed in parallel locally at the trial site prior to enrollment, but at least CPS per local testing has to be available prior to enrollment.
6. Patient has not received prior cytotoxic or targeted therapy.
7. Patient has not had a prior complete esophagogastric tumor resection.
8. Patient has a ECOG ≤ 1.
9. Patient must have life expectancy of at least 12 weeks
10. Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last study treatment if it is in the core treatment phase or for at least 3 months after last study treatment occurred in the maintenance phase. Male patients must refrain from donating sperm during this same period. Male patients with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy.
11. Patient has a body weight > 30 kg
12. Patient has adequate hematological, hepatic and renal function as indicated by the following parameters:

    1. Leukocytes ≥ 3,000/µL, platelets ≥ 100,000/µL without transfusion, absolute neutrophil count (ANC) ≥ 1,500/µL without granulocyte colony-stimulating factor support, hemoglobin ≥ 90 g/L (9 g/dL) - Patients may be transfused to meet this criterion.
    2. Bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate transaminase and alanine transaminase ≤ 2.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN
    3. Serum creatinine ≤ 1.5 x ULN, or glomerular filtration rate > 45 mL/min (calculated using the Cockcroft-Gault formula)
    4. Serum albumin ≥ 25 g/L (2.5 g/dL)
    5. For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN; for patients receiving therapeutic anticoagulation: stable anticoagulant regimen
13. Patient has no human immunodeficiency virus (HIV) infection. NOTE: Patient with infection is eligible if he/she meets all the following criteria:

    1. CD4 count is ≥350 cells/µL, viral load is undetectable, and not taking prohibited cytochrome (CYP)-interacting medications
    2. Probable long-term survival with HIV if cancer were not present
    3. Stable on a highly active antiretroviral therapy (HAART) regimen for ≥4 weeks and willing to adhere to their HAART regimen with minimal overlapping toxicity and drug-drug interactions with the experimental agents in this study
    4. HIV is not multi-drug resistant
    5. Taking medication and/or receiving antiretroviral therapy that does not interact or have overlapping toxicities with the study medication

Exclusion Criteria:

1. Patient has known hypersensitivity to any component of the durvalumab formulation as well as a known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein.
2. Patient has any known contraindication (including hypersensitivity) to docetaxel, 5-FU, leucovorin (calcium folinate), or oxaliplatin. In cases of pernicious anemia or other anemias due to vitamin B 12 deficiency, folinic acid (Leucovorin) is contraindicated and trial inclusion is not possible or only possible after compensation the anaemic status.
3. Patient has a known dihydropyrimidine dehydrogenase (DPD) deficiency. Patients with reduced DPD activity (CPIC activity score of 1.0-1.5) might participate in the study and receive a reduced dosage of 5-FU.
4. Patient has active or history of autoimmune disease including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

   NOTE: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, or controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible based on consultation with the sponsor's medical monitor. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all following conditions are met:
   * Rash must cover < 10% of body surface area.
   * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
   * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
5. Patient had a prior allogeneic bone marrow transplantation or prior solid organ transplantation.
6. Patient has a history of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, idiopathic pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.

   NOTE: History of radiation pneumonitis within the radiation field (fibrosis) is permitted.
7. Patient has active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to enrollment) or hepatitis C infection NOTE: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
8. Patient has active tuberculosis.
9. Patient has uncontrolled tumor-related pain (Patients requiring pain medication must be on a stable regimen at study entry.)
10. Patient received an administration of a live, attenuated vaccine within four weeks prior to start of enrollment, or anticipation that such a live attenuated vaccine will be required during the study or within 30 days after the last dose of durvalumab.
11. Patient had a prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibodies.
12. Patient had a treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within four weeks or five half-lives of the drug, whichever is longer, prior to study enrollment.
13. Patient had a treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to initiation of study treatment. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed

    1. Intranasal, inhaled, topical steroids or local steroid injections (e.g. intra articular injection)
    2. Systemic corticosteroids at physiologic dose not to exceed 10mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g. CT premedication)
14. Patient has a significant cardiovascular disease, such as cardiac disease (New York Heart Association Class II or greater), myocardial infarction or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmias, or unstable angina.
15. Patient has a clinically significant valvular defect.
16. Patient has a history of malignancy other than EGA within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g. 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
17. Patient has peripheral polyneuropathy ≥ NCI CTCAE grade 2.
18. Patient has uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN).
19. Patient has a serious infection requiring oral or IV antibiotics within 14 days prior to study enrollment.
20. Patient has chronic inflammatory bowel disease.
21. Patient has clinically significant active gastrointestinal bleeding.
22. Patient underwent major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment.
23. Patient has evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the study medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results.
24. Patient participated in another interventional clinical study ≤ 30 days prior to study enrollment or participation in such a study at the same time as this study.
25. Patient has taken an investigational drug within 28 days prior to initiation of study drug.
26. Female patients, who are pregnant or breast feeding or planning to become pregnant within and 6 months after the end of treatment. Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical and pathological complete response (cCR/pCR) | 8 weeks after completion of core treatment
  Rate of clinical and pathological complete response rate at time of endoscopic re-evaluation (at the end of the core study treatment) according to Becker criteria and investigator-based RECIST v1.1 assessment as well as endoscopic response criteria similar to the Japanese Gastric Cancer Association Guideline

SECONDARY OUTCOMES:
Rate of cCR/pCR (long term follow up) | 1, 2 and 3 years after start of treatment
  Rate of cCR/pCR at 1, 2 and 3 years after start of treatment (long term follow up)
Subgroup analysis of cCR/pCR | 8 weeks after completion of core treatment and after 1 year
  Subgroup analysis of cCR/pCR rate at time of endoscopic re-evaluation and after 1 year according to following characteristics: MSI high, PD-L1 CPS>1 and PD-L1 CPS>5 and especially acc. to CPS ≥10 or <10
Rate of salvage surgery | up to 48 months
  Rate of salvage surgery
Mortality | 90 days, 12 months after start of treatment
  90-day as well as 1-year mortality after start of treatment in non-surgery population and population with salvage surgery
Determination of the sites of tumor relapse | up to 48 months
  Determination of the sites of tumor relapse
Safety Endpoints | up to 20 months
  Incidence of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) as assessed during treatment and until 90 days after the last dose of study drug
  * Severity of adverse events by CTCAE v5.0 grade
  * Relationship of adverse events to the durvalumab, chemotherapy and/or radiation
  * Frequency of clinically significant abnormal laboratory parameters to CTCAE (Common Terminology Criteria for Adverse Events)

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Institut für Klinische Krebsforschung IKF GmbH; Thorsten Götze, Prof. Dr., Principal Investigator — Institute of Clinical Cancer Research, University Cancer Center (UCT) Frankfurt Krankenhaus Nordwest
Locations (22):
- Germany (22):
  - Klinikum St. Marien Kommunalunternehmen - Anstalt des öffentlichen Rechts der Stadt Amberg, Amberg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Charite Univeristätsmedizin Berlin, Berlin
  - Universitätsklinikum Brandenburg an der Havel Medizinische Hochschule Brandenburg, Brandenburg
  - Krankenhaus St. Joseph-Stift GmbH, Bremen
  - Klinikum Darmstadt GmbH, Darmstadt
  - Kliniken Essen Mitte Klinik für Internistische Onkologie und Hämatologie, Essen
  - Institute of Clinical Cancer Research, University Cancer Center (UCT) Frankfurt Krankenhaus Nordwest, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Halle (Saale) Universitätsklinik und Poliklinik für Innere Medizin I, Halle
  - Universitätsklinikum Heidelberg, RadioOnkologie & Strahlentherapie, Heidelberg
  - St. Elisabeth Gruppe GmbH, St. Anna Hospital Herne, Herne
  - Klinikverbund Allgäu gGmbH, Kempten
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - ÜBAG - Medizinisches Versorgungszentrum Dr. Vehling-Kaiser GmbH, Landshut
  - Klinikum Ludwigshafen gGmbH, Ludwigshafen
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie GEHO, Münster
  - Kreiskliniken Reutlingen GmbH Klinikum am Steinberg Reutlingen Ermstalklinik, Bad Urach, Reutlingen
  - Leopoldina-Krankenhaus Medizinische Klinik II, Schweinfurt
  - Klinikum Mutterhaus Trier, Trier
  - Klinikum Wolfsburg, Wolfsburg

IPD SHARING:
Plan to Share IPD: No